CLINICAL TRIAL: NCT05328739
Title: The Effect of Planned Homecare According to Orem on the Self-care Agency and Care Burden in Patients With Primary Brain Tumors and Caregivers: A Randomized Controlled Trial
Brief Title: The Effect of Home Care Planned According to Orem in Patients With Primary Brain Tumor and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Derya Dağdelen, Lecturer, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019/179
Record Dates: First submitted 2021-11-06; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Primary Brain Tumor; Caregiver Burden; Self Care
Keywords: caregiver burden; primary brain tumor; home care; self care agency
MeSH Terms: conditions — Brain Neoplasms; Caregiver Burden | interventions — Home Care Services

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home care group (Experimental): The home care program included education, counseling and nursing care to determine and meet the self-care/dependant care needs of patients and caregivers at home after brain surgery.
  At preoperative period (PRP) an average of 90-120 minutes of training was given to both the patient and the caregiver until the patient was discharged. At this stage, the training was carried out in order to prepare the patient and caregiver for the transition to home. At postoperative period (POP) two home visits were made within the first month following the discharge, planned for education, counseling and nursing care. The first home visit was made in the first week after discharge (10-18 days after surgery), and the second home visit was made 30-40 days after surgery. Then, in the home visits made once in the 2nd, 3rd and 4th months.No home visits were made between the 4th-month attempt and the 6th month, but telephone counseling was provided when necessary. Home visits ranged from 60 to 120 minutes.
  Interventions: Other: home care
- Control group (No Intervention): The patient received routine care in the hospital until discharge. Three home visits were made to collect the data of patients and caregivers in the 1st and 3rd and 6th months of POP after discharge, but no intervention was made. The visits took about 30-45 minutes.

INTERVENTIONS:
Other: home care — home care program
  Arms: Home care group

SUMMARY:
This study was conducted to evaluate the effect of home care planned according to Orem on self-care agency and care burden in brain tumor patients and their caregivers. The study was performed with patients who underwent surgery for a brain tumor and their caregivers in the neurosurgery clinic of a tertiary hospital. Ethical committee approval, institutional permission, patients and their caregiver verbal and written consent were obtained. According to Orem's nursing theory, home care practice combining education, counseling and nursing care started with pre-operative education in the hospital for the patients and caregivers in the intervention group and continued at home with 5 home visits in a 6-month period. Self-Care Agency Scale, MD Anderson Symptom Inventory Brain Tumor-Turkish Form and Caregiver Burden Scale were used as measurement tools in the study.The value of p<0.05 was accepted statistically significant in the data analyses.

DETAILED DESCRIPTION:
In this randomized controlled experimental study, it was aimed to determine the effect of home care planned according to Orem on self-care agency and care burden in brain tumor patients and their caregivers. The study was performed with patients who underwent surgery for a brain tumor and their caregivers in the neurosurgery clinic of a tertiary hospital. Ethical committee approval, institutional permission, patients and their caregiver verbal and written consent were obtained. According to Orem's nursing theory, home care practice combining education, counseling and nursing care started with pre-operative education in the hospital for the patients and caregivers in the intervention group and continued at home with 5 home visits in a 6-month period. Self-Care Agency Scale, MD Anderson Symptom Inventory Brain Tumor-Turkish Form and Caregiver Burden Scale were used as measurement tools in the study. In addition, measurement tools used in patients and caregivers were applied to an average of 6 month: before surgery preoperative assessment at hospital (Time 1), after surgery 1st month at home (Time 2) after surgery 3rd month at home (Time 3) and after surgery 6th month at home (Time 4). Data were analyzed with descriptive statistics, two-way analysis of variance. Bonferroni correction was applied when comparing the main effects and comparisons between categorical variables and groups were evaluated with Fisher's exact test, p<.05 value was considered statistically significant.

ELIGIBILITY:
inclusion criteria for patient;

* living within the borders of the region,
* being over 18 years old,
* being at least literate, being able to communicate in Turkish,
* being oriented to person, place and time, not having hearing and speaking problems,
* having primar brain tumor (glial or meningeal) surgery,
* taking part in grade I, II, III
* and having Karnovsky Performance Scale (KPS) score above 50 points.

exclusion criteria for patient;

* being under the age of 18,
* illiterate, unable to communicate in Turkish,
* being diagnosed with a neurological and psychiatric disorder that may affect the cognitive status,
* not being oriented to the person, place and time, having hearing and speaking problems,
* having surgery for a metastatic brain tumor,
* having surgery for a pituitary adenoma, to have undergone emergency surgery, to have a biopsy,
* to be in grade IV,
* to have a KPS score below 50 points.

Criteria for terminating the research process;

* wanting to leave the research process,
* meeting one of the criteria for exclusion from the sample after the surgery,
* spending the home care and follow-up process in another province, and/or not being able to reach the individual.

inclusion criteria for caregiver;

* being over the age of 18,
* being literate, being able to communicate in Turkish, and not having hearing and speaking problems,
* caring for a patient who had primary brain tumor surgery.

exclusion criteria for caregiver ;

* being under the age of 18,
* illiterate, unable to communicate in Turkish,
* being diagnosed with a neurological or psychiatric disorder that may affect the cognitive status,
* and having hearing and speech problems.

Criteria for terminating the research process;

* wanting to leave the research process,
* meeting one of the criteria for exclusion from the sample after the surgery,
* spending the home care and follow-up process in another province, and/or not being able to reach the individual.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Self-Care Agency Scale (SCAS) Mean Score | An average of 6 month: preoperative assessment before surgery at hospital (Time 1), after surgery 1st month at home (Time 2) after surgery 3rd month at home (Time 3) and after surgery 6th month at home (Time 4).
  SCAS: in order to evaluate the self-care agency of patients and caregiver each measurement was performed before the intervention at the time. The lowest score is 35, the highest score is 140. The highest score shows the greatest degree of self-care agency.Change= preoperative assessment before surgery at hospital (Time 1), after surgery 1st month at home (Time 2) after surgery 3rd month at home (Time 3). and after surgery 6th month at home (Time 4).
MD Anderson Symptom Inventory Brain Tumor-Turkish Form (MDA-BTSETr ) Mean Score | An average of 6 month: preoperative assessment before surgery at hospital (Time 1), after surgery 1st month at home (Time 2) after surgery 3rd month at home (Time 3) and after surgery 6th month at home (Time 4).
  MDA-BTSETr: in order to evaluate the symptoms and the impact of the symptoms on the lives of patients, each measurement was performed before the intervention at the time. The inventory consists of two parts that evaluate the symptoms and the interference of the individual's life. In the first part of the inventory, individuals are asked to rate the severity of each symptom in the last 24 hours between 0-10 (0: no symptom, 10: the most severe level of the symptom experienced). In the second part, individuals are asked to rate how much their symptoms interfere with their lives, from 0 to 10 (0: not interfered, 10: completely interfered).Change= preoperative assessment before surgery at hospital (Time 1), after surgery 1st month at home (Time 2) after surgery 3rd month at home (Time 3). and after surgery 6th month at home (Time 4).
Caregiver Burden Scale (CBS) Mean Score | An average of 6 month: preoperative assessment before surgery at hospital (Time 1), after surgery 1st month at home (Time 2) after surgery 3rd month at home (Time 3) and after surgery 6th month at home (Time 4).
  CBS: in order to evaluate the care burden of individuals who care for patients who have undergone primary brain tumor surgery, each measurement was performed before the intervention at the time. The lowest score that can be obtained from the scale is 0, the highest score is 88, and an increasing score indicates an increase in the burden of care.Change= preoperative assessment before surgery at hospital (Time 1), after surgery 1st month at home (Time 2) after surgery 3rd month at home (Time 3). and after surgery 6th month at home (Time 4).

SECONDARY OUTCOMES:
Karnofsky Performance Scale (KPS) Mean Score | An average of 6 month: preoperative assessment before surgery at hospital (Time 1), after surgery 1st month at home (Time 2) after surgery 3rd month at home (Time 3) and after surgery 6th month at home (Time 4).
  KPS allows to determine the individual and medical care needs of the patient, to obtain information about symptom severity and level of function at work and home. It is scored between 0-100. The loss of function from normal function (100) to death (0) based on the functional status of the individual. Change= preoperative assessment before surgery at hospital (Time 1), after surgery 1st month at home (Time 2) after surgery 3rd month at home (Time 3). and after surgery 6th month at home (Time 4).

CONTACTS AND LOCATIONS:
Overall Officials: Derya Dağdelen, PhD, Principal Investigator — TC Erciyes Universty
Locations (1):
- Erciyes University Faculty of Health Science, Kayseri, Eyalet/Yerleşke, Turkey (Türkiye)

REFERENCES:
- [Derived] Dagdelen D, Zincir H. Effects of dependent care theory-based post-surgical home care intervention on self-care, symptoms, and caregiver burden in patients with primary brain tumor and their caregivers: a randomized controlled trial. Support Care Cancer. 2024 Apr 18;32(5):296. doi: 10.1007/s00520-024-08488-1. PMID 38635060